CLINICAL TRIAL: NCT03361033
Title: Components of Social Functioning in Survivors of Pediatric Brain Tumors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: SOCFUN; NCI-2021-05595 (Registry Identifier: NCI)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Brain Tumor, Pediatric; Medulloblastoma, Pediatric
Keywords: Survivorship; Social Functioning; Social Outcomes
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Social Adjustment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medulloblastoma: Participants who are survivors of pediatric medulloblastoma and who meet eligibility criteria will be approached for their consent to participate in this study. Observational data will be collected through the administration of standard psychological questionnaires. If the participant consents, their parents, teachers and best friends will also be asked to complete questionnaires. In addition, participants will complete an online daily diary assessment of their social interactions for seven days.
- Other Brain Tumors: Participants who are survivors of other pediatric brain tumors (excluding medulloblastoma and craniopharyngioma), who have not been treated with craniospinal irradiation (CSI), and who meet eligibility criteria will be approached for their consent to participate in this study. Observational data will be collected through the administration of standard psychological questionnaires. If the participant consents, their parents, teachers and best friends will also be asked to complete questionnaires. In addition, participants will complete an online daily diary assessment of their social interactions for seven days.

SUMMARY:
Children with brain tumors are at risk for a number of psychological late effects, including neurocognitive and social deficits. This observational study focuses on assessment of social functioning, including social-cognitive and neurocognitive abilities, in survivors of pediatric brain tumors. This study will also assess the influence of medical factors, including diagnosis and age at diagnosis, on social functioning.

PRIMARY OBJECTIVE: Examine the impact of social-cognitive and neurocognitive abilities on social functioning in survivors of pediatric brain tumors.

SECONDARY OBJECTIVE: Assess the influence of medical factors such as diagnosis and age at diagnosis on the social functioning of survivors of pediatric brain tumors.

DETAILED DESCRIPTION:
Assessment of social and neurocognitive functioning in survivors of pediatric brain tumors who are least two years post-therapy and between 8 and 12 years of age will be included. Participants will be recruited from two tumor types: 1) medulloblastoma, and 2) other brain tumors that were not treated with craniospinal irradiation. Upon enrollment, participants will complete standard psychological questionnaires used to evaluate both performance-based and self-report measures of social and neurocognitive functioning. Parents will complete questionnaires. Families will be asked for permission to contact teachers to complete additional questionnaires. Children will identify their best friend as part of their questionnaires and will be asked permission to contact this friend to complete two questionnaires. Finally, children will be asked to complete an online daily diary of social interactions for seven days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of medulloblastoma or other brain tumor
* Current age between 8 and 12 years, inclusive
* At least 2 years post-completion of therapy
* Enrolled in school full-time
* English speaking
* Cognitive and language capacity to complete measures
* Teacher inclusion: Consent received from survivor and parent to contact.
* Best Friends inclusion: (1) Consent received from survivor and parent to contact, (2) English-speaking, (3) Cognitive capacity to complete questionnaires as judged by the parent during the consent process.

Exclusion Criteria:

* Diagnosis of a genetic disorder/pre-existing neurodevelopmental condition associated with neurocognitive or social impairment (e.g., autism, Neurofibromatosis Type 1 (NF1), Down syndrome
* Homeschooled or full-time special education
* IQ less than 70 as documented in the medical record
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Other tumor cohort exclusion: (1) diagnosis of craniopharyngioma, (2) treatment history includes craniospinal irradiation (CSI).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Potential participants will be recruited from the outpatient Neuro-Oncology, Radiation Oncology, and After Completion of Therapy Clinics at St. Jude Children's Research Hospital. Children diagnosed with either a medulloblastoma or other brain tumor, between the ages of 8 and 12 years, and at least 2 years off-therapy will be eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Significant predictors of social-cognitive and neurocognitive abilities on social functioning | From enrollment through up to 7 days later
  The primary outcome is social interaction which will be assessed via a Daily Diary that documents an individual's positive and negative social interactions, averaged over 7 days. All participants will be evaluated for the primary outcome, and descriptive statistics will be estimated to characterize the sample across all measures.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Conklin, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols